CLINICAL TRIAL: NCT03997175
Title: ImmunoGarden - Effect of Modified Playground Environment on Health, Particularly Immune System
Brief Title: Effect of Modified Playground Environment on Health, Particularly Immune System
Acronym: ImmunoG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Aki Sinkkonen, University Researcher, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HelsinkiUIG1
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Atopic Disorders; Immune System Diseases
Keywords: biodiversity intervention; sand box; guidance
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Intervention Model Description: One arm received biodiversity sand and the other arm normal sand.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants nor their parents did not know the arm. Care providers did not know the group as they did not know the content of the sand box. Investigators and field assistants knew the content in each sand box but they did not know the coding of the arms when they analyzed the differences in cytokine levels. Outcomes assessors i.e. nurses who took blood samples did not know the arms nor the contents of the sand boxes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The children were in daily contact with biodiversity sand 5 days a week for two weeks.
  Interventions: Other: Biodiversity powder
- Placebo (Placebo Comparator): Children were in contact with normal but colored sand that looked as it were the biodiversity sand. All the other details were as above.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Biodiversity powder — Biodiversity sand contained biodiversity powder that contains a highly diverse and rich microbial community but no known pathogens.
  Other Names: Biodiversity sand; Biodiversity intervention
  Arms: Intervention
Other: Placebo — Sand that looks like intervention sand but does not have high biodiversity
  Other Names: Placebo sand
  Arms: Placebo

SUMMARY:
Children were exposed to biodiverse material or non-diverse material in sand pits. The two arms were compared. Immune response and bacterial markers were followed.

DETAILED DESCRIPTION:
Children of age 3-5 were randomly divided into two groups (arms). One received guidance and biodiverse material for 20 minutes each day for two weeks. The other received the a similar material and guidance but the microbial community in the material was poor in diversity. Bacterial community changes and immune system markers were analyzed and compared between the two arms. Potential changes in Interleukin 10 was the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* born in Finland
* spends daily (5 d a week) several hours in one of the daycares in which the trial was performed

Exclusion Criteria:

* medication affecting immune system function
* medication affecting microbiota
* cancer
* immune deficiency
* living on a farm
* not born in Finland

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Interleukin 10 level in blood | two weeks
  The difference between day 0 and a follow up day in intervention

SECONDARY OUTCOMES:
changes in microbiota | two weeks
  all potential changes in bacterial profile are measured on skin and stool samples
changes in interleukin 17 levels | two weeks
  all measured changes in interleukin 17 levels
changes in tgf-beta levels | two weeks
  change in tgf-beta levels
ratio il-10 / il-17 | two weeks
  potential changes in the ratio of these two citokines
long-term changes in microbiota | four weeks
  potential changes that last for four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, ph d, Principal Investigator — University of Helsinki
Locations (1):
- Helsinki University, Lahti, Kanta-Häme, Finland

IPD SHARING:
Plan to Share IPD: Undecided
The local ethical committee and the law in Finland retricts the sharing of information that could lead to distinguishing a study participant. Microbial information is considered to faciliation the identification of study participants. Microbial information will be partly shared to public databases (sequences).